CLINICAL TRIAL: NCT04822597
Title: Optimizing Topical Pain Control for Breast Cancer Patients Undergoing Pre-operative Radiotracer Injection for Sentinel Lymph Node Mapping
Brief Title: Pain Control for Breast Cancer Patients Receiving Injection of Radioactive Tracer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-0261; A539713 (Other: UW Madison); SMPH/SURGERY/SURG ONC (Other: UW Madison); UW20164 (Other: UWCCC); Protocol Version 3/2022 (Other: UW Madison); 2T32CA090217-16 (NIH)
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Sentinel Lymph Node; Breast Neoplasms; Breast Cancer Female
Keywords: Sentinel Lymph Node Biopsy; Sentinel Lymph Node Mapping; Radioactive Tracer Injection; Nuclear Medicine; Radiocolloid Injection
MeSH Terms: conditions — Breast Neoplasms | interventions — Ice

STUDY DESIGN:
Intervention Model Description: There will be four separate treatment arms. Participants have equal chances of being assigned to any of the four arms.
Who Masked: Outcomes Assessor
Masking Description: Data will be analyzed with intervention arms masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Ice Pack (Active Comparator): Ice will be placed on the breast prior to radioactive tracer injection (usual treatment)
  Interventions: Other: Ice pack
- Lidocaine Patch (Experimental): A lidocaine patch (4% topical) will be placed on the breast for at least one hour prior to radioactive tracer injection
  Interventions: Drug: Lidocaine patch
- Buzzy(R) (Experimental): A vibrating distraction device (Buzzy(R)) and ice will be placed on the breast prior to radioactive tracer injection.
  Interventions: Device: Buzzy(R); Other: Ice pack
- Lidocaine Patch and Buzzy(R) (Experimental): A lidocaine patch (4% topical) will be placed on the breast for at least one hour prior to radioactive tracer injection. This will be removed and a vibrating distraction device (Buzzy(R)) and ice will be placed on the breast just prior to radioactive tracer injection.
  Interventions: Drug: Lidocaine patch; Device: Buzzy(R); Other: Ice pack

INTERVENTIONS:
Drug: Lidocaine patch — Lidocaine is a local anesthetic.
  Other Names: topical lidocaine 4%
  Arms: Lidocaine Patch; Lidocaine Patch and Buzzy(R)
Device: Buzzy(R) — Buzzy provides non-invasive pain relief by vibrating and cooling the skin which distracts from pain sensations.
  Other Names: vibrating distraction device; therapeutic vibrator
  Arms: Buzzy(R); Lidocaine Patch and Buzzy(R)
Other: Ice pack — Ice cools the skin and can provide some numbing for pain.
  Other Names: ice; coolant
  Arms: Buzzy(R); Ice Pack; Lidocaine Patch and Buzzy(R)

SUMMARY:
The purpose of this study is to compare the effectiveness four different pain treatments for the injection of radioactive tracer that women with breast cancer receive for sentinel lymph node biopsies.

This study will include women who have been diagnosed with breast cancer and who will be undergoing sentinel lymph node biopsy with a standard injection of radioactive tracer before surgery.

A participant's active participation will take place on two separate occasions. In the first occasion, a participant will complete a brief pain assessment on the day of enrollment. The rest of a participant's active participation will take place on one day (the day of surgery) and last approximately 20 minutes, after which active participation will end.

DETAILED DESCRIPTION:
Primary Objective: To test the effectiveness of four alternative approaches to topical anesthesia on pain associated with radiotracer injection for women diagnosed with breast cancer undergoing sentinel lymph node mapping.

Secondary Objectives:

1. To assess patient satisfaction with pain control modality for radiotracer injection.
2. To identify barriers to implementation of the different pain control interventions.

ELIGIBILITY:
Inclusion Criteria:

* greater than or equal to 18 years of age
* biopsy proven breast cancer
* standard radiotracer injection (intradermal injection in the upper outer quadrant of the involved breast)
* radiotracer injection occurs on the same day as sentinel lymph node surgery

Exclusion Criteria:

* males
* pregnancy
* local anesthetic allergy or active use of the following medications:

  * Abametapir (risk X)
  * Conivaptan (risk X)
  * Fusidic Acid (risk X)
  * Idelalisib (risk X)
  * Mifepristone (risk D)
  * Stiripentol (risk D)
  * Amiodarone (risk C)
  * Dofetilide (risk C)
  * Dronedarone (risk C)
  * Ibutilide (risk C)
  * Sotalol (risk C)
  * Vernakalant (risk C)
* Non-English speaking/reading
* Unable to provide informed consent
* Unable to participate with surveys
* Undergoing radiotracer injection the day prior to surgery or intra-operatively at the time of initial surgical scheduling

  * If patients are initially scheduled for same-day preoperative injection, complete all enrollment procedures (including randomization), and surgery is re-scheduled for a day prior to surgery or for intra-operative injection, they will be excluded if:

    * randomized to a lidocaine patch arm (Arms C or D)
    * re-scheduled for an intra-operative injection • Planned non-standard radiotracer injection site

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather B Neuman, MD, Principal Investigator — University of Wisconsin Madison School of Medicine and Public Health
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from the UW Hospital and Clinics were enrolled from April 2021 to January 2022.
Period: Overall Study
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Started | 44 | 39 | 44 | 40
On Treatment As Assigned | 44 | 37 | 35 | 34
Off Treatment As Assigned | 44 | 37 | 35 | 34
Analyzed With Intent to Treat | 43 | 37 | 42 | 38
Completed | 43 | 37 | 42 | 38
Not Completed | 1 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Subject withdrawn after enrollment | 0 | 1 | 0 | 1
Not completed — Surgery Re-scheduled, missed by study team | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R) | Total
Number analyzed (Participants) | 44 | 39 | 44 | 40 | 167
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 2 | 2 | 2 | 2 | 8
  40-49 years | 6 | 7 | 7 | 7 | 27
  50-59 years | 6 | 14 | 11 | 10 | 41
  60-69 years | 16 | 10 | 14 | 11 | 51
  70-79 years | 14 | 4 | 9 | 10 | 37
  80-89 years | 0 | 2 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 39 | 44 | 40 | 167
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 41 | 38 | 43 | 40 | 162
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 2 | 0 | 1 | 4
  White | 42 | 37 | 44 | 37 | 160
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 44 | 39 | 44 | 40 | 167

OUTCOME MEASURES:

1. Primary Outcome: Median Post-Procedural Pain Score
Description: Post-procedural pain score on the Wong-Baker FACES scale. Scale from 0-10 with 0 being "no pain" and 10 being "worst pain".
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
score on a scale | 2 [2 to 6] | 2 [2 to 4] | 4 [2 to 6] | 4 [2 to 4]

2. Secondary Outcome: Short Form McGill Sensory Pain Score
Description: Sensory pain score out of 33 with 0 being "no pain" and 33 being severe sensory pain
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
score on a scale | 1 [0 to 3] | 1 [0 to 3] | 2 [0 to 5] | 2 [0 to 3]

3. Secondary Outcome: Short Form McGill Affective Pain Score
Description: Affective pain score out of 12 with 0 being "no pain" and 12 being severe affective pain
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
score on a scale | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 2] | 0 [0 to 0]

4. Secondary Outcome: Short Form McGill VAS Pain Score
Description: Visual analog scale pain score out of 100 with zero being "no pain" and 100 being "worst possible pain"
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
score on a scale | 24 [14 to 66] | 28 [19 to 39] | 27 [16 to 53] | 33 [14 to 50]

5. Secondary Outcome: Short Form McGill Combined Pain Score
Description: Combination of outcomes 2-3. Additive total score between 0 and 45 with zero being "no pain" and 45 being "severe pain"
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
score on a scale | 4 [1 to 9] | 3 [1 to 7] | 6 [2 to 9] | 3 [2 to 6]

6. Secondary Outcome: Degree of Participant Satisfaction With Attention Paid to Complaints as Reported by Number of Participants Who Report Satisfied or Very Satisfied
Description: 1-6 scale with 1 being "very satisfied" and 6 being "very dissatisfied". Reported are the number of participants satisfied or very satisfied.
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Count of Participants; unit: Participants
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
Participants | 42 | 37 | 42 | 37

7. Secondary Outcome: Degree of Participant Satisfaction With Care Provided During Injection as Reported by Number of Participants Who Report Satisfied or Very Satisfied
Description: as for outcome 6
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Count of Participants; unit: Participants
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
Participants | 42 | 37 | 42 | 37

8. Secondary Outcome: Degree of Participant Satisfaction With Pain Control as Reported by Number of Participants Who Report Satisfied or Very Satisfied
Description: as for outcome 6
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Count of Participants; unit: Participants
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
Participants | 33 | 33 | 36 | 36

9. Secondary Outcome: Degree of Anxiety During the Injection as Measured by Number of Participants Moderately Anxious
Description: 1-4 scale with 1 being "very anxious" and 4 being "not at all anxious", reported here are the number of participants rating anxiety at 2 or "moderate".
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Count of Participants; unit: Participants
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
Participants | 33 | 24 | 32 | 25

10. Secondary Outcome: Recommendation of Pain Control Modality as Measured by Number of Participants Who Answered "Yes"
Description: "Yes", "No", "Not sure" with option for free response
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Measure: Count of Participants; unit: Participants
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
Participants | 31 | 31 | 35 | 35

11. Secondary Outcome: Provider Perceived Ease of Administration
Description: 7 point single ease question to rate ease of a task. 1 being "very difficult" and 7 being "very easy". This is the provider's perception of the how easy the intervention was to administer.
Time Frame: Day of surgery (last of two study visits), assessed within 30 minutes of radioactive tracer injection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
score on a scale | 7 [6 to 7] | 6 [5 to 7] | 7 [6 to 7] | 6 [5 to 7]

12. Secondary Outcome: Provider Perceived Participant Pain
Description: 11 point numeric rating scale for perceived pain of others. 0 being "no pain" and 7-10 being "severe pain".
Time Frame: Day of surgery, assessed within 30 minutes of radioactive tracer injection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 43 | 37 | 42 | 38
score on a scale | 3 [3 to 6] | 3 [2 to 5] | 4 [3 to 5] | 3 [2 to 5]

13. Secondary Outcome: Provider Rank Ordering Ease of Use of Interventions
Description: End of study survey to compare providers' perceived usability of intervention. Rank ordering of interventions 1-4 with 1 being "easiest to administer" and 4 being "hardest to administer".
Time Frame: Assessed after last participant off study (up to 12.5 months)
Population: There were 8 providers surveyed to rank the ease of use of the interventions, they were not consented as the IRB considered them 'study team members'
Measure: Count of Participants; unit: Participants
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants
  1 - easiest to administer | 1 | 0 | 7 | 0
  2 | 7 | 0 | 1 | 0
  3 | 0 | 8 | 0 | 0
  4 - hardest to administer | 0 | 0 | 0 | 8

14. Secondary Outcome: Provider Rank Ordering Perceived Efficacy of Interventions
Description: End of study survey to compare providers' perceived efficacy of intervention. Rank ordering of interventions 1-4 with 1 being "best pain control" and 4 being "least pain control".
Time Frame: Assessed after last participant off study (up to 12.5 months)
Population: There were 8 providers that were not consented to the study because the IRB considered the 'study team members'
Measure: Count of Participants; unit: Participants
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
Number analyzed (Participants) | 8 | 8 | 8 | 8
Participants
  1 - best pain control | 2 | 2 | 0 | 4
  2 | 2 | 4 | 2 | 0
  3 | 2 | 1 | 1 | 4
  4 - worst pain control | 2 | 1 | 5 | 0

ADVERSE EVENTS:
Time Frame: Day of surgery (last of two study visits), assessed within 3 hours of radioactive tracer injection
Arm/Group | Ice Pack | Buzzy(R) | Lidocaine Patch | Lidocaine Patch and Buzzy(R)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/39 | 0/44 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/39 | 0/44 | 0/40
Other Adverse Events (participants affected / at risk) | 0/44 | 0/39 | 0/44 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT04822597/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT04822597/ICF_000.pdf